CLINICAL TRIAL: NCT06344143
Title: Detecting Mild Autonomous Cortisol Secretion in Patients With Adrenal Incidentaloma
Acronym: MACS
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-324
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mild Autonomous Cortisol Secretion (MACS)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Various labs and imaging tests — Dexamethasone Suppression Test, Adrenocorticotropic Hormone (ACTH), Salivary Cortisol Levels, Vasopressin Stimulation test, Fasting Glucose, Fasting Insulin, Complete Metabolic Panel (CMP), Gamma-glutamyl transferase (GGT), Sex Hormone Binding Globulin, Cat scan of abdomen/Pelvis, Whole body dual energy x-ray absorptiometry (DXA) scan, Ultrasound Fibroscan Transient Elastography

SUMMARY:
The aim of the proposed study is to estimate the incidence of Mild Autonomous Cortisol Secretion (MACS) in patients with Adrenal Incidentaloma (AI) and evaluate the available diagnostic tests to determine the most sensitive and specific combination of tests for assessing MACS from adrenal adenoma for prediction of the phenotype associated with cortisol excess. As well as following the patients for 4 years and see if anything changes.

DETAILED DESCRIPTION:
Mild Autonomous cortisol secretion (MACS) is defined as the hypersecretion of cortisol by the adrenal glands, independent of Adrenocorticotropic Hormone (ACTH) regulation. MACS can be a challenging diagnosis for clinicians to make. It is commonly associated with adrenal incidentalomas (AI), the incidental finding of adrenal gland masses on cross-sectional imaging. There are a variety of adverse clinical conditions associated with MACS, including central obesity, hypertension, impaired fasting glucose due to insulin resistance, and dyslipidemia, which together comprise the "metabolic syndrome," as well as type 2 diabetes mellitus, cardiovascular disease, osteoporosis with vertebral fractures, and early mortality. Androulakis et al. concluded that patients with AI, even without hypertension, diabetes, and/or dyslipidemia, may still have adverse cardiovascular outcomes, possibly due to increased insulin resistance and endothelial dysfunction linked to subtle cortisol excess. There is also a reported association of non-alcoholic fatty liver disease (NAFLD), an increasingly significant cause of morbidity and mortality, with the metabolic syndrome and diabetes, as well as hypercortisolism. However, the link between MACS and NAFLD has not been well delineated, nor has the effect of treatment with MACS on NAFLD been explored.

Given the findings cited above, there may be benefit in treating patients with AI and MACS with medical therapy. Therefore, identifying those individuals who have the metabolic syndrome or its components, bone disease, NAFLD, or increased cardiovascular risk related to excess cortisol secretion is essential but difficult.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 18 years and older.
2. Presence of adrenal incidentaloma by cat scan (CT) or magnetic resonance imaging (MRI) examination.
3. 1-mg Dexamethasone suppression test cortisol ≤ 5 μg/dL with adequate dexamethasone level.

Exclusion Criteria:

1. 1-mg Dexamethasone suppression test cortisol > 5 μg/dL with adequate dexamethasone level. Patients who fail to suppress below this level will be considered to have Cushing's syndrome and will be referred for appropriate treatment.
2. Current or recent (3 months) history of use of glucocorticoid medication (including joint injections of steroids).
3. History of uncontrolled hypertension or history of hypertension with more than 2 medications.
4. History of uncontrolled type 2 Diabetes Mellitus or history of diabetes mellitus with A1c>7.5.
5. Known History of osteoporosis
6. Documented Clinical Cushing's disease.
7. Clinical suspicion of adrenal carcinoma.
8. History of alcohol abuse/dependence.
9. History of cirrhosis of liver.
10. History of hepatitis B or C infection regardless of treatment.
11. History of type 1 diabetes.
12. History of hemochromatosis.
13. History of autoimmune hepatitis.
14. History of Wilson's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from Endocrinology patients who have previously undergone dexamethasone suppression testing for Adrenal Incidentaloma (AI) or have been diagnosed with AI and have been seen at the Endocrinology and Metabolism institute (EMI). They will be identified from review the laboratory database and clinical records. All subjects with a dexamethasone suppression test <5 micrograms/dL will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate best diagnostic test(s) | 5 years
  To evaluate and determine the most sensitive and specific combination of tests for assessing mild autonomous cortisol secreting (MACS) from adrenal adenoma for prediction of the phenotype associated with cortisol excess. Study team will measure cortisol in serum, cortisol in saliva, cortisol in urine, vasopressin stimulation test, 1 mg dexamethasone stimulation test (DST) and a 2 mg DST, Adrenocorticotropic Hormone test (ACTH) and (dehydroepiandrosterone sulfate test) DHEAS. With this, a diagnosis of MACS can be determined. To determine the sensitivity of each the area under the curve (AUC) will be compared with the standard test which is 1 mg DST.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Correa, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No